CLINICAL TRIAL: NCT01478269
Title: Prognosis Of Patients With Aggressive B-Cell Lymphoma, Treated With Rituximab+Anthracycline Regimen (ProDLBCL)
Brief Title: Prognosis Of Patients With Aggressive B-Cell Lymphoma, Treated With Rituximab+Anthracycline Regimen
Acronym: ProDLBCL
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: IIL_ProDLBCL
Record Dates: First submitted 2011-10-12; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: B-Cell Lymphomas
Keywords: Aggressive B-cell lymphoma; R-CHOP
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cases of aggressive B-cell lymphoma: Cases of aggressive B-cell lymphoma diagnosed between 2001 to 2007 in Italy

SUMMARY:
This study is a retrospective analysis of an homogeneous population of patients with aggressive B-cell lymphoma and treated upfront with R-CHOP or R-CHOP like regimens to reassess the prognostic factors and hopefully to identify more accurate prognostic subgroups with a clinical and therapeutical relevance.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed newly diagnosed aggressive B-cell lymphoma according to the current World Health Organisation Classification, from 2001 to 2007.
2. Any stage of disease.
3. Treatment with R-CHOP or R-CHOP like regimens (+/- transplant).
4. Age at least 18 years.
5. Availability of tissue biopsy at diagnosis for a possible centralized revision.
6. Availability of data on clinical involvement, laboratory, treatment and follow up.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases of aggressive B-cell lymphoma diagnosed between 2001 to 2007 in Italy
Sampling Method: Non-Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2009-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Federico, MD, Study Director — Oncologia II Azienda Ospedaliera Universitaria di Modena; Stefano Luminari, MD, Principal Investigator — Oncologia II Azienda Ospedaliera Universitaria di Modena
Locations (39):
- Brazil (4):
  - Hemocentro-Unicamp, Campinas
  - Centro Medico, Santa Isabel
  - Centro Paulista de Oncologia, São Paulo
  - Santa Casa Medical School, São Paulo
- Italy (35):
  - Clinica Ematologica Policlinico Carreggi, Florence, Firenze
  - Ematologia e Trapianto IRCCS, Istituto Nazionale dei Tumori, Milan, Milano
  - A.O.SS. Biagio, Antonio e Cesare Arrigo, Alessandria
  - Centro di riferimento Oncologico Oncologia Medica A, Aviano (Pordenone)
  - USC Ematologia e Trapianto di Midollo Osseo Ospedali Riuniti di Bergamo, Bergamo
  - Presidio Ospedaliero A.Perrino - Divisione di Ematologia, Brindisi
  - U.O. di Oncologia Ospedale di Circolo di Busto Arsizio, Busto Arsizio
  - Ospedale Civile, Camposanpiero (PD)
  - A.O.Pugliese Ciaccio Diviisone di Ematologia, Catanzaro
  - Presidio Ospedaliero Annunziata U.O.C. di Ematologia, Cosenza
  - Ematologia 1 Ospedale S. Martino, Genova
  - Oncologia Medica B e C IST Genova, Genova
  - Ospedale Felettino, La Spezia
  - Ospedale Madonna delle grazie U.O. Ematologia, Matera
  - A O Papardo, Messina
  - Azienda Ospedaliero Universitaria Policlinico Gaetano Martino, Messina
  - Oncologia Medica 3 Istituto Nazionale dei Tumori di Milano, Milan
  - Osp. San Carlo Borromeo Divisione di Oncologia Medica, Milan
  - Ospedale Maggiore IRCCS-Dipartimento di Ematologia, Milan
  - Centro Oncologico Modenese, Modena
  - A.O. Maggiore della Carità S.C.D.U. Ematologia, Novara
  - A.O. di Padova Divisione di Oncologia Medica, Padua
  - Casa di cura La Maddalena Unita' di Ematologia, Palermo
  - Div. di Ematologia e TMO AOU Policlinico Giaccone di Palermo, Palermo
  - A O Universitaria di Parma, Parma
  - Ospedale Civile G.da Saliceto - UOA Ematologia, Piacenza
  - Azienda Ospedaliero Universitaria Pisana U.O. Ematologia, Pisa
  - AO Bianchi Melacrino Morelli UO Ematologia, Reggio Calabria
  - AO Arcispedale S.Maria Nuova Ematologia, Reggio Emilia
  - Ospedale Oncologico regionale CROB, Rionero in Vulture (PZ)
  - Dipartimento di biotecnologie cellulari ed ematologia Ospedale Umberto I - La Sapienza, Roma
  - Policlinico A. Gemelli Università Cattolica del Sacro Cuore, Roma
  - Clinica Humanitas, Rozzano (MI)
  - A.O.San Giovanni Battista, Torino
  - U.O. Oncologia Azienda ULSS7 P.O. di Vittorio Veneto, Vittorio Veneto